CLINICAL TRIAL: NCT05802836
Title: Dynamics of the Anti-factor VIII Antibody Signature During Treatment With Emicizumab
Acronym: NAVIGATE
Status: Recruiting | Type: Observational
Sponsor: Christoph Königs (Other)
Collaborators: Roche Pharma AG (Industry); Chugai Pharma Germany GmbH (Unknown)
Responsible Party: Sponsor-Investigator, Christoph Königs, Principal Investigator, Head of molecular and clinical Haemostasis, Goethe University
Organization: Goethe University (Other)
Other Study IDs: ML44394; DRKS00031196 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2023-03-06; First posted 2023-04-07 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Severe Hemophilia A; Severe Hemophilia A With Inhibitor; Severe Hemophilia A Without Inhibitor
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inhibitor negative, FVIII on demand or regularly: Patients with severe hemophilia A receiving emicizumab therapy which are negative for factor VIII Inhibitor (including patients post ITI) and are receiving factor VIII therapy either on demand or regularly,
  Interventions: Other: no interventions
- Inhibitor positive, FVIII therapy regularly (ITI): Patients with severe hemophilia A receiving emicizumab therapy which are positive for factor VIII Inhibitor and are receiving regularly factor VIII therapy (ITI)
  Interventions: Other: no interventions
- Inhibitor positive, no FVIII therapy: Patients with severe hemophilia A receiving emicizumab therapy which are positive for factor VIII Inhibitor and are receiving no factor VIII therapy
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no intervention, only 3 different patients groups

SUMMARY:
The goal of this observational study is to learn about the changes of antibodies and inhibitors against the coagulation factor VIII in patients with severe hemophilia A receiving emicizumab therapy. No additional visits or procedures are planned. Patients in this study will continue to receive their routine care and analysis will be done from left over samples from routine visits.

ELIGIBILITY:
Inclusion Criteria:

* Severe congenital hemophilia A (CHA)
* Treatment with emicizumab irrespective of any other treatment
* Informed consent

Exclusion Criteria:

* No therapy with emicizumab
* Immunosuppressive therapy
* HIV-infection with CD4 (cluster of differentiation 4) cells <200/µl

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to recruit 100 patients with severe hemophilia A from 15 study sites in germany.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
FVIII inhibitor development in inhibitor negative subjects | 3 years
  Rate of FVIII inhibitor development during three years of emicizumab prophylaxis in inhibitor negative subjects. Assessed with Bethesda Assay (BU/ml). Number of patients who develop an FVIII inhibitor within the study period, but were FVIII inhibitor negative at start of the study.
FVIII antibody development in inhibitor negative subjects | 3 years
  Rate of FVIII antibody development during three years of emicizumab prophylaxis in inhibitor negative subjects. FVIII anti drug antibody (ADA) is assessed by FVIII specific ELISA (OD=Optical Density). Number of patients who develop an FVIII antibody (ADA) within the study period, but were FVIII inhibitor negative at start of the study.
FVIII inhibitor disappearance in inhibitor positive subjects | 3 years
  Rate of FVIII inhibitor disappearance during three years of emicizumab prophylaxis in inhibitor positive subjects. Assessed with Bethesda Assay (BU/ml). Number of patients who loose an FVIII inhibitor within the study period, but were FVIII inhibitor positive at start of the study.
FVIII antibody disappearance in inhibitor positive subjects | 3 years
  Rate of FVIII antibody disappearance during three years of emicizumab prophylaxis in inhibitor positive subjects. FVIII anti drug antibody (ADA) is assessed by FVIII specific ELISA (OD=Optical Density). Number of patients who develop an FVIII antibody within the study period, but were FVIII inhibitor positive at start of the study.

SECONDARY OUTCOMES:
Anti-FVIII inhibitor development | 3 years
  Anti-FVIII inhibitor development (median BU/ml) over time. Assessed with Bethesda Assay (BU/ml). Description of inhibitor development in the different patient groups within the study period. Cut off is 0,6 BU/ml.
Anti-FVIII antibody development | 3 years
  Anti-FVIII antibody development (median arbitrary units, OD) over time. Description of antibody development in the different patient groups within the study period.
Time to negative inhibitor titers | 3 years
  Time to negative inhibitor titers. Assessed with Bethesda Assay (BU/ml). Description of the Time (days) observed for FVIII inhibitor disappearance within the study period in the patient groups. Cut off for inhibitor titer is 0,6 BU/ml.
Treatment of bleeds | 3 years
  Description of the use of FVIII and/or Bypassing agents treatment in addition to Emicizumab treatment in case of bleeds.
Response to treatment | 3 years
  Classification of bleeds as Effective, Partially Effective, Ineffective. Defined as: Effective: Bleeding episode responded to the usual number of injections or dose of FVIII as expected by the treating physician; Partially Effective: The bleeding episode responded with a higher number of injections and/or dose as expected by the treating physician; Ineffective: Routine failure to control hemostasis or hemostatic control required additional agents
Quality of the antibody response (FVIII epitopes) | 3 years
  Description of the location of FVIII epitopes over time, assessed by epitope mapping technique (ELISA)
Quality of the antibody response (IgG subclasses) | 3 years
  Description of a potential immune response over time, assessed by IgG subclass determination (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Koenigs, PD Dr. Dr, Principal Investigator — Goethe University
Locations (1):
- University Hospital Frankfurt, Goethe University, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No